CLINICAL TRIAL: NCT02822742
Title: A Phase III, Open-label, Single-arm, Multi-center Study Assessing the Safety and Efficacy of DE-117 Ophthalmic Solution in Subjects With Primary Open-angle Glaucoma or Ocular Hypertension Who Are Non-/Low-responders to Latanoprost Ophthalmic Solution: FUJI Study
Brief Title: A Study Assessing the Safety and Efficacy of DE-117 in Subjects With POAG or OH Who Are Non-/Low-responders to Latanoprost: FUJI Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01171506
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Primary Open Angle Glaucoma or Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DE-117 ophthalmic solution and Latanoprost (Other): DE-117 is Experimental. Latanoprost is Active Comparator.
  Interventions: Drug: DE-117 ophthalmic solution; Drug: Latanoprost ophthalmic solution 0.005%

INTERVENTIONS:
Drug: DE-117 ophthalmic solution
Drug: Latanoprost ophthalmic solution 0.005%

SUMMARY:
The purposes of this study are to investigate the effect of intraocular pressure lowering efficacy and safety of DE-117 ophthalmic solution in subjects with primary open-angle glaucoma or ocular hypertension who are non-/low-responders to latanoprost ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma or ocular hypertension

Exclusion Criteria:

* Patients at risk of progression of visual field loss
* Patients with severe visual field defect
* Patients with any diseases that preclude participation in this study for safety reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure | Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Tokyo, Japan

REFERENCES:
- [Derived] Aihara M, Ropo A, Lu F, Kawata H, Iwata A, Odani-Kawabata N, Shams N. Intraocular pressure-lowering effect of omidenepag isopropyl in latanoprost non-/low-responder patients with primary open-angle glaucoma or ocular hypertension: the FUJI study. Jpn J Ophthalmol. 2020 Jul;64(4):398-406. doi: 10.1007/s10384-020-00748-x. Epub 2020 Jun 22. PMID 32572719